CLINICAL TRIAL: NCT03808974
Title: An Educational Video to Improve Patient Comprehension of Midurethral Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Felicia Lane (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor-Investigator, Felicia Lane, Professor, Urogynecology Division Director, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20184707
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Stress Urinary Incontinence; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Urinary Incontinence, Stress; Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will be shown an educational video
  Interventions: Other: Educational video
- Control (Active Comparator): The control group will be given an educational leaflet
  Interventions: Other: Educational leaflet

INTERVENTIONS:
Other: Educational video — Short educational video describing the mid-urethral sling procedure
  Arms: Intervention
Other: Educational leaflet — Standard educational leaflet describing the mid-urethral sling procedure
  Arms: Control

SUMMARY:
The purpose of this research project is to test the effectiveness of a previsit educational video designed to help women understand the risks and benefits of a midurethral sling for treatment of stress urinary incontinence. A total of 38 participants will be recruited from both the Urogynecology pre-operative clinic of the university of California, Irvine Medical Center and the Urogynecology pre-operative clinic at Kaiser Permanente, Anaheim and Orange County. Participants will be randomized either to watch a 10 minute educational video (intervention group) or read a standard handout describing the midurethral sling (control group). Participants will then complete their pre-operative visit in the usual fashion. Participants will complete a pre- and post- intervention knowledge questionnaire to assess the primary outcome (change in knowledge before and after intervention). Participants will repeat the knowledge questionnaire and complete validated questionnaires for satisfaction with decision scale and decision regret at 2 and 6 weeks post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for a mid-urethral sling for stress urinary incontinence with a urogynecology provider at a participating hospital

Exclusion Criteria:

* < 18 years of age
* Non-English speaking or requiring interpreter assistance
* Presence of cognitive dysfunction
* Women receiving a repeat midurethral sling (not primary)
* Women with a history of pelvic mesh complication (erosion, pain, history of mesh excision)
* Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Patient knowledge questionnaire (investigator-created) | 6 weeks
  The change in participant knowledge as measured with a patient knowledge questionnaire. This questionnaire was created by the study investigators and piloted by physicians within our institutions. It was submitted to and approved by our IRB for use in this study. This is a 15-point questionnaire (true/false/unknown answer choices) in which 1 point is given for each correct response and 0 points given for incorrect or unanswered questions (minimum score: 0/15, maximum score: 15/15). The questions pertain to the risks, benefits, and procedure of the mid-urethral sling surgery. Higher scores indicate better participant knowledge. A subscale of mesh-related questions will also be examined. This subscale reports the participant knowledge pertaining to complications and procedural knowledge specific to the use of mesh in the mid-urethral sling. The scale of this subset ranges from 0/5 to 5/5, with higher scores indicating greater participant knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, MD, Study Director — University of California, Irvine
Locations (1):
- University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeney SES, Whitcomb EL, Ihara J, Guaderrama N, Mukhtar F, Heliker BD. A Randomized Controlled Trial Evaluating the Effect of an Educational Video on Patient Understanding of Midurethral Sling. Female Pelvic Med Reconstr Surg. 2022 Mar 1;28(3):e73-e79. doi: 10.1097/SPV.0000000000001154. PMID 35272337